CLINICAL TRIAL: NCT05912972
Title: Development and Management of Registry in Patients With Gynecologic Cancer in Korea
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-Yeol Park, MD, PhD, Professor, Asan Medical Center
Other Study IDs: 2022-1412
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Cervical Cancer; Endometrial Cancer; Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cervical cancer: No interventions
  Interventions: Other: Patient registry
- Endometrial cancer: No interventions
  Interventions: Other: Patient registry
- Ovarian cancer, Fallopian tube cancer, Peritoneal cancer: No interventions
  Interventions: Other: Patient registry

INTERVENTIONS:
Other: Patient registry — Clinical data, specific procedures and treatments will follow the Institutional standard operative procedures

SUMMARY:
The goal of this observational study is to identify and analyze the characteristics, treatment trends, prognostic factors and survival prognosis of Korean gynecologic cancer patients. Ultimately, the final goal is to contribute to the development of safe surgical methods and treatment for gynecologic cancer to improve survival rates.

DETAILED DESCRIPTION:
Cervical cancer, endometrial cancer, and ovarian cancer represent gynecologic cancers. There are many open issues that need to be addressed, specifically the surgical method, disease recurrence and survival outcome in the so called "real world" setting. The aim of this observational study is to collect both retrospective and prospective medical information of gynecologic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years or older
* Written informed consent (prospective cohort)
* Confirmed diagnosis of cervical cancer, endometrial cancer or ovarian cancer

Exclusion Criteria:

* Unconfirmed diagnosis of cervical cancer, endometrial cancer or ovarian cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gynecologic cancer undergoing treatment
Sampling Method: Probability Sample
Enrollment: 13500 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2027-10-21 (Estimated); Study Completion 2027-10-21 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Analyzed for all patients as time from diagnosis to death as a result of any cause, stratified according to baseline characteristics, surgical methods, and treatment

SECONDARY OUTCOMES:
Progression-free survival | 5 years
  Analyzed for all patients, as time from diagnosis to progression of disease or death as a result of any cause, stratified according to baseline characteristics, surgical methods, and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Yeol Park, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea